CLINICAL TRIAL: NCT05380245
Title: Pharmacokinetic Drug-Drug Interaction Study of Voriconazole With Clarithromycin.
Brief Title: Drug-Drug Interaction Study of Voriconazole With Clarithromycin.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abdul Wali Khan University Mardan (Other)
Responsible Party: Principal Investigator, Dr. Yasar Shah, Associate Professor, Abdul Wali Khan University Mardan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Dir/A&R/AWKUM/2018/1408-25; AWKUM-16002974 (Other: Abdul Wali Khan University Mardan,Pakistan)
Record Dates: First submitted 2022-04-03; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Voriconazole (Voriz); Clarithromycin (CLRM); Washout period; Randomized; Pharmacokinetic drug-drug interaction (PK-DDI); Clinical significance
MeSH Terms: interventions — Voriconazole; Clarithromycin

STUDY DESIGN:
Intervention Model Description: A single dose, randomized, crossover, open-labeled and two sequence study with a two-week washout period, evaluated the impact of clarithromycin on the pharmacokinetics (PK) profile of voriconazole Pakistani healthy male volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Voriconazole (alone), then Voriconazole + Clarithromycin. (Experimental): On Day-1, Group-A participants first received Voriconazole (alone) (Dose: 400mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral). After a washout period of two weeks. Then, on Day-16 they received Voriconazole (Dose: 400mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral) along with Clarithromycin (Name of medication of Intervention Formulation: Tablet Klaricid, Dose: 500mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral).
  Interventions: Drug: Voriconazole 200 mg x 2 Tablets; Drug: Clarithromycin 500 mg x 1Tablets
- Treatment Voriconazole + Clarithromycin, then Voriconazole (alone). (Experimental): On Day-1, Group-B participants first received Voriconazole (Dose: 400mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral) along with Clarithromycin (Name of medication of Intervention Formulation: Tablet Klaricid, Dose: 500mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral).After a washout period of two weeks. Then, on Day-16 they received Voriconazole (alone) (Dose: 400mg, Dosage form: Tablet, Frequency: Once (OD), Duration of administration: Single Dose, Kind of administration: Oral).
  Interventions: Drug: Voriconazole 200 mg x 2 Tablets; Drug: Clarithromycin 500 mg x 1Tablets

INTERVENTIONS:
Drug: Voriconazole 200 mg x 2 Tablets — Name of medication of Reference Formulation: Tablets Voriconazole Vfend®, 200 mg by Pfizer, Inc. (USA), (Batch No: 00005505; Mfg. date 09/2016).
  Other Names: Vfend®
Drug: Clarithromycin 500 mg x 1Tablets — Name of medication of Intervention Formulation: Tablet Klaricid, 500 mg by Abbott, Lab Pvt. Ltd. (Karachi, Pakistan), Batch No: 81573XU; Mfg. date 10/2017.
  Other Names: klaricid®

SUMMARY:
The current study evaluated the Pharmacokinetic (PK) drug-drug interaction (PK-DDI) of voriconazole with clarithromycin in healthy male volunteers. The drug interaction study was designed as a single oral dose, open-label, crossover, and randomized trial. In the first phase of the study, the principal investigator developed a high-performance-liquid chromatography (HPLC) method and validation according to standard ICH guidelines for the quantification of voriconazole in the biological matrix. During the second step, Enrolled volunteers were divided randomly into group A and group B by the "permuted block randomization" technique. Then, voriconazole either alone (2 x 200mg, tab, P/O) or in combination with clarithromycin (Voriconazole 2 x 200mg, tab + clarithromycin 500mg, tab, P/O) was administered to enrolled volunteers in two sequences. Finally, sample collection was carried out and blood samples were collected at specified time periods (i.e., 0.0 (pre-dose), 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, and 24 hours) in EDTA or heparinized tubes from the enrolled human volunteers. Further processing of the sample was done for extractions and subsequent analysis with the developed analytical method.

DETAILED DESCRIPTION:
Study Design and Ethical Approval: The drug interaction study was designed as a single oral dose, open-label, randomized, cross-over study of healthy volunteers. The ethical approval of the protocol was taken from the Advanced Studies and Research Board (ASRB) of the Pharmacy department, Abdul Wali Khan University, Mardan before initiation. This study followed the "ethical principles of the Helsinki declaration for medical research involving human subjects" and "good clinical practice guidelines". The clinical trial of this study followed the guidelines of CONSORT. Written consent was obtained from all included volunteers in the DDI study. The study was comprised of two treatment sequences with a two-week washout period

Randomization and Drug administration: Enrolled volunteers were divided randomly into Group A and Group B by the "permuted block randomization" technique. Computed the volunteer data into an excel sheet and applied a RAND* function; selected two groups (G-A and G-B) sized, finally assigned 6 participants in each study group for two (Voriz (alone) or Voriz + CLRM) intervention arms, for the execution of block randomization. A balance (1:1) was acquired across both intervention arms through this randomization technique. Treatment drugs were administered to enrolled volunteers in two sequences,

Sequence-I: In the first phase, group-A volunteers on day-1 received oral voriconazole (2 x 200mg, tab, P/O) while group-B volunteers received oral clarithromycin (500mg, tab, P/O) along with voriconazole (2 x 200mg, tab, P/O). A two-week wash-out period was allocated that started on day-2 to day-15 for avoiding the carry-over effect.

Sequence-II: On day-16, the second phase of the trial was conducted in which group-A volunteers received voriconazole (2 x 200mg, tab, P/O) along with clarithromycin (500mg, tab, P/O) while group-B volunteers received Voriz (2 x 200mg, tab, P/O) only. Voriconazole and clarithromycin were administered to the overnight fasted volunteers corresponding to the sequences. All volunteers took the medication with a glass of water (250mL). On day-1 and 16 (treatment days), standard breakfast and lunch were served two and six hours after drug administration to all volunteers, respectively.

ELIGIBILITY:
Inclusion Criteria:

• Male Pakistani volunteers in good health aged 18-35 years were enrolled as participants in this study.

The selection was based on:

* A complete detailed medical history,
* Clinical examination,
* Voriconazole hypersensitivity test,
* Evaluation of various biochemical tests like Blood Glucose Level, Hemoglobin (Hb) Level, Serum Glutamic-Pyruvic Transaminase (SGPT) Or Alanine Amino Transferase and Aspartate (ALT and AST, respectively) Level, Urine Test, Albumin to Creatinine Ratio (ACR) Test, Glomerular Filtration Rate (GFR) Level, etc.

Exclusion Criteria:

* Those volunteers were having a history of voriconazole hypersensitivity reaction were excluded from the study.
* Deviation from normal values in the biochemical test report was excluded from the study.
* Having any pathology like chronic renal disease, and hepatic impairment was excluded from the study.
* Having any cardiovascular, gastrointestinal tract, and hematopoietic disorders were excluded from the study.
* Alcohol addicted, smokers and volunteers who cannot sign the permission consent form were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of voriconazole | At "Day 1" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose and At "Day 16" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose.
  Determine the Plasma Concentration particularly the Maximum Plasma Concentration (Cmax) of voriconazole either alone or co-administration with clarithromycin.
Area under the Plasma Concentration versus Time Curve (AUC) of voriconazole | At "Day 1" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose and At "Day 16" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose.
  Determine the Area under the Plasma Concentration versus Time Curve (AUC) of voriconazole either alone or co-administration with clarithromycin.

SECONDARY OUTCOMES:
Maximum Time to Reach (Cmax) of voriconazole (Tmax) | At "Day 1" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose and At "Day 16" Pre-dose, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour post-dose.
  Tmax of voriconazole either alone or co-administration with clarithromycin.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mehwish Mushtaq, MPhil, Principal Investigator — Abdul Wali Khan University Mardan (AWKUM), Pakistan / Metrics Research Organization CRO, Pakistan.; Dr. Yasar Shah, Ph.D., Study Director — Abdul Wali Khan University Mardan (AWKUM), Pakistan.
Locations (1):
- Medical Dispensary, Abdul Wali Khan University Mardan, Pakistan., Mardan, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
To keep the confidentiality of the study participants, however, data would be made available to the Ethics Committee of the institute upon requirement.

REFERENCES:
- [Derived] Mushtaq M, Fatima K, Ahmad A, Mohamed Ibrahim O, Faheem M, Shah Y. Pharmacokinetic interaction of voriconazole and clarithromycin in Pakistani healthy male volunteers: a single dose, randomized, crossover, open-label study. Front Pharmacol. 2023 Jun 9;14:1134803. doi: 10.3389/fphar.2023.1134803. eCollection 2023. PMID 37361220

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05380245/Prot_SAP_ICF_000.pdf